CLINICAL TRIAL: NCT00313391
Title: The Effects of Risperdal Consta on Health Care Utilization Costs in Chronically Ill Schizophrenic Patients
Brief Title: Risperdal Consta and Health Care Utilization in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Janssen, L.P. - Investigator Initiated Studies Program (Unknown)
Responsible Party: Dragan Bugarski-Kirola, MD, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 731-2005
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: Risperdal Consta

SUMMARY:
The purpose of this study is to determine if Risperdal Consta will affect the healthcare utilization costs in chronically ill schizophrenic patients with multiple admissions to the psychiatric hospital compared to the previous utilization costs under standard oral treatment of any atypical antipsychotic. We hypothesize that higher Risperdal Consta acquisition costs can be offset by reduction in total medical utilization costs, such as hospitalizations, ER visits, unscheduled outpatient visits or incarcerations due to worsening of psychotic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of schizophrenia or schizoaffective disorder
* 4 or more admissions to psychiatric hospital in past year, OR minimum of 2 hospital admissions and at least 2 incarcerations in the previous year
* Medicaid recipient
* Patients requiring concomitant non-antipsychotic psychotropic medication (mood stabilizing, antidepressants, anxiolytics)

Exclusion Criteria:

* Past or current psychiatric disorder, other than schizophrenia or schizoaffective disorder
* Drug or alcohol dependence
* Serious, unstable medical illness or any acute medical condition
* Pregnant or lactating females
* Prior Risperdal Consta treatment
* Non-English speaking

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Dates: Start 2005-12; Primary Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragana Bugarski-Kirola, MD, Principal Investigator — Emory University
Locations (1):
- Grady Hospital, Atlanta, Georgia, United States